CLINICAL TRIAL: NCT02406352
Title: Development and Application of a Multispectral Digital Colposcope and Probe Algorithm for Detection of Cervical Intraepithelial Neoplasia
Brief Title: Multispectral Digital Colposcope With Probe for Detection of Cervical Intraepithelial Neoplasia
Acronym: MDCwProbe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brookdale University Hospital Medical Center (Other)
Responsible Party: Principal Investigator, Michele Follen, Chair of Department of Obstetrics and Gynecology, Brookdale University Hospital Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-35
Record Dates: First submitted 2015-03-16; First posted 2015-04-02 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Carcinoma in Situ of Uterine Cervix; Cervical Intraepithelial Neoplasias; High Grade Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

ARMS (1):
- Routine colposcopy and MDC with probe (Experimental): The intervention which consists of obtaining cervical images with the MDC and spectroscopic data with the probe will be applied to all participants who agreed to participate in the study during their visit for a colposcopy exam or treatment with a LEEP procedure. A control biopsy will also be obtained from patients who agree to provide it. The control biopsy is a biopsy of cervical tissue that does not appear to have atypical changes when observed through a standard of care colposcope.
  Interventions: Device: Multispectral Digital Colposcope with probe

INTERVENTIONS:
Device: Multispectral Digital Colposcope with probe — Cervical images will be obtained with the Multispectral Digital Colposcope. Spectroscopic data will be obtained with the probe from eligible patients who provided consent to participate in the study.
  The standard of care for research participants will not change.

SUMMARY:
Although cervical cancer is a preventable cancer, every year more than one-quarter of a million women die worldwide from this disease. Internationally and nationally, cervical cancer is a disease that affects predominantly women who are poor and who live in resource poor settings. With the device the investigators are developing, known as the Multispectral Digital Colposcope with probe, our goal is to make detection of precancerous cervical lesions easier for the patient and for her provider. For the patient, our goal is to reduce the number of clinical visits needed to obtain a diagnosis and treatment and consequently to reduce the resulting fear and anxiety which usually accompanies an abnormal Pap smear. For the provider and the health care system, our goal is to obtain a more accurate diagnosis than the currently available diagnostic methods.

DETAILED DESCRIPTION:
The multispectral digital colposcope (MDC) is a specialized lightsource and imaging device mounted on a custom-made colposcope that acquires a sequence of fluorescence images. This version of the MDC incorporates an upgraded light source, and updates the firmware and the user interface. This results in shorter acquisition times and improved image and spectrum quality control. The MDC also consists of a point probe that is used to take detailed light measurements (call spectroscopy) from smaller regions of the cervix. The goal of the study is to see whether the MDC can perform better than standard methods in detecting cancerous or pre-cancerous abnormalities of the cervix.

Study subjects will be swabbed for detection and typing of the Human Papilloma Virus (HPV). After vinegar is applied on the cervix as per usual colposcopy practice, the MDC will then be used to take a sequence of images of the cervix. Next 2-4 readings will be taken from the cervix using the point probe.

This data will be used to train, test and validate an algorithm specific to the MDC. The ability of the algorithm to detect cervical intraepithelial neoplasia will be compared to standard clinical care (colposcopy).

The MDC images and pathology results will be compared to the spectroscopy data from the MDC probe. The investigators will determine if spectroscopy has equal sensitivity to colposcopy for detecting high grade lesions.

ELIGIBILITY:
Inclusion Criteria:

* Women who are at least 18 years old
* Are not pregnant (negative urine test) or breastfeeding
* Referred for colposcopy or LEEP treatment
* Can provide written informed consent

Exclusion Criteria:

* Women who do not meet the inclusion criteria
* Women who have had a hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Detection of precancerous cervical lesions or cervical cancer | At point of care for colposcopy or treatment with LEEP (5 minutes).
  Eligible patients who are referred to the colposcopy clinic for a diagnosis following an abnormal Pap smear will be asked to participate in the study. All participating women will receive their standard of care colposcopy as usual. In addition to their routine care, the MDC with probe will also be used to collect images of the cervix and spectroscopic measurements with the probe. All measurements will be compared with the biopsies obtained. The MDC with probe will not be used to determine from where the biopsies need to be obtained. One or two additional biopsies will be obtained from tissue that appears to be unaffected. These will be the control biopsies. Patients may refuse to provide the additional biopsies which are not part of the standard of care.
  Patients scheduled for a treatment with the Loop Electrosurgical Excision Procedure (LEEP) will be asked for consent to obtain one or two biopsies prior to the LEEP procedure, but after anesthesia has been applied.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, MD, PhD, Principal Investigator — Brookdale University Hospital and Medical Center
Locations (1):
- Brookdale University Hospital and Medical Center, Brooklyn, New York, United States